CLINICAL TRIAL: NCT00542906
Title: Functional Organization of Somatosensory Responses in the Secondary Somatosensitive Area (SII) and Insula : an fMRI Study
Brief Title: Functional Organization of Somatosensory Responses in the Secondary Somatosensitive Area and Insula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint Etienne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0701023; 2007-A00328-45; DGS 2007-0273
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: healthy volunteers; Somatosensory stimuli; fMRI; second somatosensory area; insular cortex; functional anatomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): healthy volunteers
  Interventions: Other: localization

INTERVENTIONS:
Other: localization — localization of the several types of somatosensory stimuli

SUMMARY:
The implication of the second somatosensory area (SII) and the insular cortex in the processing of somatosensory inputs is now well established. However the functional anatomy of these areas hidden in the depth of the sylvian scissure remain mostly unknown.

The aim of this fMRI study is to determine the functional cartography of SII and insula. The localization of responses to different somatosensory stimuli (slight touch, warm, cold, heat pain and arthrokinesia) applied on the left hand of 25 healthy volunteers, will be compared.

DETAILED DESCRIPTION:
Aims : Demonstrate that localization of the several types of somatosensory stimuli is different into SII and into insula. If possible, we'll determine a functional cartography of these areas.

ELIGIBILITY:
Inclusion Criteria:

* 25 healthy volunteers will be included ranging in age from 18 to 50 years
* contraception needed for women
* right handed
* All the subjects have to give their written informed consent.

Exclusion Criteria:

* pregnancy
* neurological or psychiatric disease
* drugs taken <12h before fMRI
* contra-indications to fMRI : pacemaker, clip, metallic device
* Refusing to be informed of the presence of a cerebral abnormality, detected during MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Comparison of euclidian distances between the centroids of clusters activations for the different types of stimulations into SII and insula. | one day

SECONDARY OUTCOMES:
Determine the Talairach coordinates of the centroids of clusters of activations for the different types of somatosensory stimuli into SII and insula | one day

CONTACTS AND LOCATIONS:
Overall Officials: Laure Mazzola, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Service de Neurologie - CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Mazzola L, Isnard J, Mauguiere F. Somatosensory and pain responses to stimulation of the second somatosensory area (SII) in humans. A comparison with SI and insular responses. Cereb Cortex. 2006 Jul;16(7):960-8. doi: 10.1093/cercor/bhj038. Epub 2005 Sep 21. PMID 16177270
- [Background] Peyron R, Schneider F, Faillenot I, Convers P, Barral FG, Garcia-Larrea L, Laurent B. An fMRI study of cortical representation of mechanical allodynia in patients with neuropathic pain. Neurology. 2004 Nov 23;63(10):1838-46. doi: 10.1212/01.wnl.0000144177.61125.85. PMID 15557499